CLINICAL TRIAL: NCT03263052
Title: An Evaluation of Converting Elderly Kidney Transplant Recipients From Tacrolimus to Envarsus to Limit Neurological Adverse Events and Improve Quality of Life
Brief Title: Converting Elderly Kidney Transplant Recipients From Tacrolimus to Envarsus to Limit Neurological AE and Improve QOL
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Patricia West-Thielke, Director of Clinical Research, University of Illinois at Chicago
Other Study IDs: 2017-0400
Record Dates: First submitted 2017-08-22; First posted 2017-08-28 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Disorder Related to Renal Transplantation
Keywords: kidney transplant; immunosuppression; tacrolimus XR; elderly; quality of life; neurological adverse events
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Tacrolimus XR
  Interventions: Drug: Tacrolimus XR (Envarsus)

INTERVENTIONS:
Drug: Tacrolimus XR (Envarsus) — Elderly patients (age 60 or older) on tacrolimus experiencing neurological AEs (tremor, insomnia, vertigo, photophobia, mood disturbances, or headache) presumably from tacrolimus immediate-release or tacrolimus XL will be converted to Envarsus. This conversion will be based on the Envarsus package insert which is a 20% reduction in total daily dose and is taken once a day. The conversion from Astagraf to Envarsus will be a 36% reduction.

SUMMARY:
This study will investigate whether converting patients from FDA approved immediate-release tacrolimus to FDA approved extended release tacrolimus (Envarsus) reduces neurological side-effects, improves quality of life, and enhances adherence. A select group of elderly (> 60 years of age) patients, who are especially sensitive to tacrolimus-related adverse (AEs) effects, will be provided the opportunity to convert to Envarsus with this study.

DETAILED DESCRIPTION:
Tacrolimus (Prograf) is a calcineurin inhibitor that is widely used in all types of solid organ transplants. However, one of the major limitations in using tacrolimus are the adverse effects that significantly reduce a transplant recipient's quality-of-life (QOL). These QOL reducing AEs associated with tacrolimus include post-transplant diabetes mellitus, neurotoxicity, diarrhea, nephrotoxicity, and alopecia. A recent open-label, multicenter, prospective phase 3b study showed that Envarsus significantly reduced tremors and improved quality of life when compared to tacrolimus. It is postulated that the mechanism behind tremor reduction occurs as a result of lower Cmax tacrolimus concentrations with the new Envarsus formulation. Given its ability for tremor improvement, it would be beneficial to investigate whether conversion from tacrolimus to Envarsus can improve other neurological AEs such as insomnia vertigo, photophobia, mood disturbances, or headache. In particular, the elderly are especially sensitive to tacrolimus-related AEs and may benefit from tacrolimus to Envarsus conversion. Further, it is useful to understand the cost effectiveness of converting to Envarsus in this patient population.

Study duration: 35 days per subject until a total of 40 subjects are enrolled. Patients will have a total of 4 visits.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a recipient of a living donor or deceased donor kidney only transplant
2. Subject is > 60 years of age
3. Subject reports neurological AEs from tacrolimus that include one or more of the following: insomnia, vertigo, photophobia, mood disturbances, tremor, and/or headache.
4. Patients must be able to understand English and provide written informed consent
5. Patients receiving a stable dose (i.e., no dose adjustments) of immediate-release tacrolimus (Prograf) or extended-release tacrolimus (Astagraf) for a minimum of 4-7 days at screening
6. Patients with a screening tacrolimus trough level of 3-12 ng/mL, measured between Day -7 to 0
7. The patient is not scheduled to begin any new medication that could interfere with tacrolimus blood levels, including prescription and over-the-counter medications, herbal or food supplements (including grapefruit and pomegranate products)
8. Patients must be willing to commit to and comply with the schedule of study visits

Exclusion Criteria:

1. Multi-organ transplant
2. Subjects not taking tacrolimus post-transplant
3. Documented Parkinson's disease or dementia
4. Known cause of neurological symptoms other than tacrolimus
5. Patients with significant visual and hearing impairments affecting their ability to complete the study requirements and assessments
6. Patients with any severe medical condition (including infection) requiring acute or chronic treatment that in the Investigator's opinion would interfere with study participation
7. Known non-adherence (defined as documentation in the patient chart of multiple missed visits and/or medication doses) which in the investigator's opinion would interfere with the objectives of the study
8. Patients who are taking any acute or chronic medications that may impact reaction time, memory, or sleep habits, based on Investigator discretion
9. Patients with any form of current drug or alcohol abuse as assessed by the Investigator

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll elderly kidney transplant recipients who are at least 60 years of age and have experienced neurological adverse events while on generic tacrolimus, Prograf, or Astagraf XL.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Quality of life (QOL) | through study completion, an average of two years
  Mean change in QOL scores from baseline to day 14 and day 28 after conversion from tacrolimus to Envarsus.
Neurological Scores | through study completion, an average of two years
  Mean change in neurological scores (including insomnia, vertigo, photophobia, mood, headache, and tremor) from baseline to day 14 and day 28 after conversion from tacrolimus to Envarsus.

SECONDARY OUTCOMES:
Tacrolimus preference | through study completion, an average of two years
  Proportion of patients preferring Envarsus compared with their previous tacrolimus formulation after 28 days of treatment
Non-adherence | through study completion, an average of two years
  Percent of patients reporting non-adherence from baseline to day 14 and 28 after conversion from tacrolimus to Envarsus.
Incremental costs | through study completion, an average of two years
  Mean incremental costs from baseline to day 28 following conversion to Envarsus.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No